CLINICAL TRIAL: NCT03640936
Title: Total IgE and Der p 1 (d1) Specific IgE in Induced Sputum in Patients With Allergic and Non-allergic Asthma
Brief Title: Total IgE (Immunoglobulin E) and Der p 1 (d1) Specific IgE in Induced Sputum in Patients With Allergic and Non-allergic Asthma
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-ASM-2014-66
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Asthma
Keywords: asthma; allergy; specific IgE
MeSH Terms: conditions — Asthma; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Supernatant of induced sputum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy: Healthy controls, without asthma or allergy (negative prick test)
  Interventions: Behavioral: Induced Sputum
- Allergic asthma: Patients with allergic asthma sensitized to Dermatophagoides pteronyssinus, tested by prick test or specific IgE
  Interventions: Behavioral: Induced Sputum
- Non-allergic asthma: Patients with asthma not sensitized to Dermatophagoides pteronyssinus, with negative prick test or specific IgE
  Interventions: Behavioral: Induced Sputum

INTERVENTIONS:
Behavioral: Induced Sputum — Total IgE and Specific IgE to Dermatophagoides pteronyssinus in Induced Sputum

SUMMARY:
Asthma is a heterogeneous disease, and specifically the phenotype of non-allergic asthma is not yet well defined. Several studies describe this group of patients as having severe asthma, persistent eosinophilia and poor therapeutic response. Among the theories being considered is the role of local IgE. Objectives: 1) To perform a pilot test to validate the measurement technique and standardize the levels of total IgE and IgE specific to Dermatophagoides pteronyssinus (d1) in the induced sputum of asthmatic patients and healthy volunteers. 2) Correlate local total IgE and specific IgE levels to d1 (sputum and peripheral blood) in patients with allergic and non-allergic asthma. 3) Describe the clinical and inflammatory characteristics of patients with allergic and non-allergic asthma.

DETAILED DESCRIPTION:
Comparative cross-sectional study. It will include 32 allergic and non-allergic asthma patients and 10 healthy volunteers. All patients will have an induced sputum, pulmonary function studies, FENO (exhaled fraction of nitric oxide), total and specific IgE measurement at d1 (the most common perennial pneumoallergen) in blood and induced sputum, as well as a prick skin test with standardized allergen extracts. Measurement of total IgE and IgE for d1 in induced sputum will be performed in the supernatant and by the ImmunoCAP (Phadia ThermoFisher Scientific) immunofluoroassay technique.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70
* Asthma according to GEMA (spanish asthma guideline)

Exclusion Criteria:

* Pregnancy
* Active smoking
* Moderate alcohol consumption
* Atopic dermatitis
* Other respiratory disease different than asthma (COPD, bronchiectasis, cystic fibrosis, pleural disease, interstitial disease)
* Treatment with steroids or inmunodepressants
* Active malignancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with asthma without evidence of allergic disease.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2015-02; Primary Completion 2017-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Levels of specific IgE | 8 months
  Detection of high levels or not of specific IgE in induced sputum

SECONDARY OUTCOMES:
Levels of total IgE | 8 months
  Detection of high levels or not of total IgE in induced sputum

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau. Carrer Mas Casanovas 90., Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Johansson SG, Bieber T, Dahl R, Friedmann PS, Lanier BQ, Lockey RF, Motala C, Ortega Martell JA, Platts-Mills TA, Ring J, Thien F, Van Cauwenberge P, Williams HC. Revised nomenclature for allergy for global use: Report of the Nomenclature Review Committee of the World Allergy Organization, October 2003. J Allergy Clin Immunol. 2004 May;113(5):832-6. doi: 10.1016/j.jaci.2003.12.591. PMID 15131563
- [Background] Wenzel SE. Asthma phenotypes: the evolution from clinical to molecular approaches. Nat Med. 2012 May 4;18(5):716-25. doi: 10.1038/nm.2678. PMID 22561835
- [Background] Crespo A, Giner J, Torrejon M, Belda A, Mateus E, Granel C, Torrego A, Ramos-Barbon D, Plaza V. Clinical and inflammatory features of asthma with dissociation between fractional exhaled nitric oxide and eosinophils in induced sputum. J Asthma. 2016 Jun;53(5):459-64. doi: 10.3109/02770903.2015.1116086. Epub 2016 Jan 19. PMID 26785727
- [Background] Rondon C, Campo P, Zambonino MA, Blanca-Lopez N, Torres MJ, Melendez L, Herrera R, Gueant-Rodriguez RM, Gueant JL, Canto G, Blanca M. Follow-up study in local allergic rhinitis shows a consistent entity not evolving to systemic allergic rhinitis. J Allergy Clin Immunol. 2014 Apr;133(4):1026-31. doi: 10.1016/j.jaci.2013.10.034. Epub 2013 Dec 13. PMID 24332860
- [Background] Baba S, Kondo K, Toma-Hirano M, Kanaya K, Suzukawa K, Ushio M, Suzukawa M, Ohta K, Yamasoba T. Local increase in IgE and class switch recombination to IgE in nasal polyps in chronic rhinosinusitis. Clin Exp Allergy. 2014;44(5):701-12. doi: 10.1111/cea.12287. PMID 24931597
- [Background] Pin I, Gibson PG, Kolendowicz R, Girgis-Gabardo A, Denburg JA, Hargreave FE, Dolovich J. Use of induced sputum cell counts to investigate airway inflammation in asthma. Thorax. 1992 Jan;47(1):25-9. doi: 10.1136/thx.47.1.25. PMID 1539140
- [Background] Margarit G, Belda J, Juarez C, Martinez C, Ramos A, Torrejon M, Granel C, Casan P, Sanchis J. [Total IgE in the sputum and serum of patients with asthma]. Allergol Immunopathol (Madr). 2005 Jan-Feb;33(1):48-53. doi: 10.1157/13070609. Spanish. PMID 15777524
- [Background] Korn S, Haasler I, Fliedner F, Becher G, Strohner P, Staatz A, Taube C, Buhl R. Monitoring free serum IgE in severe asthma patients treated with omalizumab. Respir Med. 2012 Nov;106(11):1494-500. doi: 10.1016/j.rmed.2012.07.010. Epub 2012 Aug 11. PMID 22884459
- [Background] Vega JM, Badia X, Badiola C, Lopez-Vina A, Olaguibel JM, Picado C, Sastre J, Dal-Re R; Covalair Investigator Group. Validation of the Spanish version of the Asthma Control Test (ACT). J Asthma. 2007 Dec;44(10):867-72. doi: 10.1080/02770900701752615. PMID 18097865
- [Background] Plaza Moral V; Comite Ejecutivo de GEMA. [GEMA(4.0). Guidelines for Asthma Management]. Arch Bronconeumol. 2015 Jan;51 Suppl 1:2-54. doi: 10.1016/S0300-2896(15)32812-X. Epub 2015 Nov 30. No abstract available. Spanish. PMID 26707419
- [Derived] Crespo-Lessmann A, Curto E, Mateus E, Soto L, Garcia-Moral A, Torrejon M, Belda A, Giner J, Ramos-Barbon D, Plaza V. Total and specific immunoglobulin E in induced sputum in allergic and non-allergic asthma. PLoS One. 2020 Jan 29;15(1):e0228045. doi: 10.1371/journal.pone.0228045. eCollection 2020. PMID 31995587
- See also: Spanish guideline of Asthma — http://www.gemasma.com.